CLINICAL TRIAL: NCT04204486
Title: A Multidisciplinary Evaluation on the Effects of an Exercise Intervention on Markers of Health, Wellbeing and Performance in Law Enforcement Workers
Brief Title: Health, Wellbeing and Performance in Law Enforcement Workers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13985/004
Record Dates: First submitted 2019-12-03; First posted 2019-12-19 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Musculoskeletal Pain; Cognitive Change; Occupational Stress; Inflammation
Keywords: Exercise; Strength; Source Memory; Context Memory; Inhibition; Executive Function; SOSI; Shift work; police; law enforcement; military; Oral health; Quality of Sleep; Cognition; Fitness
MeSH Terms: conditions — Musculoskeletal Pain; Occupational Stress; Inflammation; Motor Activity; Inhibition, Psychological; Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a randomised control trial. Participants will be stratified by shift pattern and by role, and will be randomised to one of three intervention arms using permuted blocks of 3 and 6.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face to face exercise intervention (Experimental): Participants will participate in face to face exercise programme delivered by a strength and conditioning coach. Sessions will last 1 hour, 3 times a week, and will be offered at the work place. The coach will register attendance in order to monitor compliance.
  Interventions: Behavioral: Exercise
- Online exercise intervention (Active Comparator): Participants will be given the same training programme as the face to face group, but via an online app. Sessions should last 1 hour and should be completed 3 times a week. Participants will be asked to post a "work-out picture" on the social platform of the app as proof that they completed their session.
  Interventions: Behavioral: Exercise
- Control (No Intervention): This group will undergo all pre and post tests, but will not receive an intervention.

INTERVENTIONS:
Behavioral: Exercise — Functional strength training, 1 hour, 3 times a week.
  Arms: Face to face exercise intervention; Online exercise intervention

SUMMARY:
This study aims to assess current health and fitness of law enforcement workers in various roles, and to evaluate the impact of an exercise intervention on markers on physical and mental wellbeing in this population.

The intervention will consist of an exercise programme specifically targeted at improving, physical fitness and reducing musculoskeletal pain. Participants will be randomised to three groups: a face to face intervention group, an online intervention group an a control group.

Self-reported physical health, musculoskeletal complaints, quality of sleep and occupational stress will be measured via questionnaires. Pre and post measures of fitness will be measured via functional strength testing and a cardiopulmonary exercise test. Pre and post cognitive function will be measured via computer-based cognitive tests and brain functional near-infrared spectroscopy (fNIRS). Systemic inflammation will be measured via hsCRP. Risk of typeII diabetes will be measured via HbA1c. Daily physical activity and quality of sleep will be measured via accelerometry and heart rate telemetry.

It is hypothesised that, upon completion of the programme, there will be an improvement in cardiovascular fitness and physical strength, reduced musculoskeletal pain, improved cognitive readiness and improved overall mental health and wellbeing.

DETAILED DESCRIPTION:
Randomisation Participants will be stratified by shift pattern and by role, and will be randomised to one of three intervention arms using permuted blocks of 3 and 6.

Self-reported information After the consent forms and PAR-Q have been signed, an Operational Police Stress Questionnaire (PSQ-Op), Impact of Events Scale (IES-R), a Leeds Sleep Evaluation (LSE) and an overall health and injury questionnaire (Nordic scale) will be sent to the officers via email using Gorilla software in December 2019.

Participants will be interviewed on the quality of their dietary intake. Trained nutrition research students will collect responses to a Food Frequency Questionnaire (FFQ) in a face to face interview.

Wearables Participants will be given wearable devices to measure their levels of physical activity during an 8-day period (full on and off shift cycle) before the intervention: the heart rate of each participant will be monitored via a Polar heart rate monitor and movement will be measured via an accelerometer worn on the non-dominant wrist (Actigraph, Pensacola, USA). Levels of physical activity, quality of sleep and heart rate variability will be processed as anonymised data on a computer. Participants will be asked to log the quality of their sleep every time they wake up from a long sleep via a Pittsburgh Sleep Quality Index (PSQI). No individuals other than the researchers will have access to the data from the wearable devices. The data will be downloaded from the device and stored in a password-protected file, on an encrypted, password-protected UCL computer in a locked cabinet. After downloading the data to the computer, the wearable device will be formatted.

Oral tests Participant oral health will be assessed on site at the respective stations in January. Oral inflammation has been shown to affect systemic health with cross-sectional evidence suggesting a negative effect on physical activity in Brazilian police. Oral health will be assessed using validated outcome measures routinely employed in both NHS dental practice and research, including: the visual assessment of inflammation of the gum edge and measurement of the depth of the gum pocket (mm) following gentle probing with a calibrated blunt probe; and tooth decay screening assessed through standard clinical methods. Together, these assessments take approximately 15 minutes.

Saliva will be analysed to investigate the effect of the physical activity intervention on the health outcomes. The researchers will collect around 5ml of saliva using standard methods by asking participants to drool into collection pots. The samples will be frozen then analysed for biomarkers related to stress and inflammation. The samples will be collected at the first and last study visits.

Physical and Cognitive tests Participants will then attend a physical screening session at the Institute of Sport, Exercise and Health (ISEH) at UCL. The session will consist of a functional strength test (triple hop, jumps to fatigue on jump mat, successful press-ups one minute, successful inverted rows in one minute). Cardiorespiratory performance will be measured via a Cardio-Pulmonary Exercise Test (CPET) on a treadmill (h/p/cosmos) using the Bruce protocol. During the CPET, Heart Rate will be monitored via a Polar heart rate monitor, and breath-by-breath analysis will be performed with a Vyair gas analyser system to collect VO2 data.

Biomarkers (hsCRP, HbA1c) will be analysed by collecting one blood capillary sample with a finger prick. The capillary is then inserted in an Eppendorf tube and inserted into a Eurolyser Cube (Eurolyser, Salsburg, Austria) to measure markers of inflammation.

Cognitive tests will be performed before and after the CPET. Participants will undergo Source & Context Memory, inhibition and SOSI tests on an encrypted computer, using the e-Prime software. The cognitive tasks will be standard-format computerised tasks that are used in e.g. studies of drug effects upon cognition, or in experiments looking at the effects of sleep deprivation, or the effects of exercise upon people's abilities to think and remember. Participants are shown pictures and words on a laptop and have to make responses using button boxes of the keyboard. The number of errors and reaction times are recorded. The tests are not stressful and no deception is involved. There are several thousands of publications in the literature that have used these or very similar procedures, and the investigators know of no case where these have caused harm to the participants.

In order to record brain activity during the cognitive tests, functional near-infrared spectroscopy (fNIRS) will be used (Shimadzu LightNIRS). An fNIRS cap placed on the participant's head records brain activity using infra-red light.

Intervention After all screening is complete, participants will be randomly allocated to one of three groups: face to face exercise program (F2F), online exercise program delivered via mobile app (APP) and control (C). The F2F group will receive three exercise training sessions, three times a week for 8 weeks, delivered in person by a strength and conditioning coach at the police station. The exercise intervention will take the format of circuit training using body weight and elastic resistance, focusing on strength endurance and core stability. The APP group will receive online instructions via an app (TeamBuilder) on how to perform the same exercise programme at home. The C group will not receive an intervention.

Behaviour change (to retain levels of physical activity during and after the intervention) will be facilitated by encouraging buddying during the exercise intervention, and by assigning points to the groups based on attendance. There will be two F2F groups and 2 APP groups (Heathrow vs Wood Green). A competitive element will be added between respective F2F and APP groups by assigning 1 point for each participant that attends the session, +2 extra points if all participants attend. Attendance will be kept by the coach for the F2F group. Participants on the APP group will be asked to take a picture of themselves after having completed each session as proof of completion. The coach will monitor compliance for both groups with at attendance spreadsheet.

Post testing After the 8-week training programme is complete, the participants will repeat the same questionnaires, wearables period, fitness tests and cognitive tests that were used in the pre-intervention testing.

Behaviour change will be assessed via a focus group after the intervention. The focus groups will be aimed at gathering feedback on the intervention and on attitudes towards exercise following the COM-B model, including participant experience and whether they felt that the intervention effectively improved their wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Working in law enforcement

Exclusion Criteria:

* Participants with any form of physical injury, neuromuscular, respiratory or cardiovascular condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in musculoskeletal pain: measured via the Nordic Scale | Change from baseline after 8 weeks
  Complaints of musculoskeletal pain, collected via a Nordic Scale. The scale runs from 0-10, where 0 is no pain at all and 10 is worst imaginable pain.
Change in upper body strength endurance (push) | Change from baseline after 8 weeks
  Numbers of pushups performed in one minute with good form (eg. not dipping the hips and using full range of motion)
Change in upper body strength endurance (pull) | Change from baseline after 8 weeks
  Numbers of inverted rows performed in one minute with good form (eg. not dipping the hips and using full range of motion)
Change in leg strength, measured via the Triple Hop test | Change from baseline after 8 weeks
  Participants perform three hops on one leg. The total distance (cm) of the three hops is recorded. The test is repeated for both legs.
Change in lower limb power | Change from baseline after 8 weeks
  Participants perform a counter-movement jump on a jump mat (Chronojump). Power (Watts) is recorded.
Change in hand grip strength | Change from baseline after 8 weeks
  Hand grip strength (Newtons) is measured with a hand-held dynamometer.
Change in Cardiovascular fitness | Change from baseline after 8 weeks
  measured via CPET test

SECONDARY OUTCOMES:
Change in simple reaction time after maximal exercise | Change from baseline after a single bout of maximal exercise (CPET)
  Measured via cognitive tests on a computer screen using the ePrime software, which require the participant to press a key on the key board after seeing a specific image. Reaction time (milliseconds) and number of errors are recorded.
Change in simple reaction time after an exercise intervention | Change from baseline after 8 weeks
  Measured via cognitive tests on a computer screen using the ePrime software, which require the participant to press a key on the key board after seeing a specific image. Reaction time (milliseconds) and number of errors are recorded.
Change in Motor Inhibition after maximal exercise | Change from baseline after a single bout of maximal exercise (CPET)
  Measured via cognitive tests on a computer screen using the ePrime software, which require participants to press a key on the keyboard every time a new image appears on the screen, except when a specific picture appears (specified in the instructions), in which case they must refrain from pressing the key. Reaction time (milliseconds) and number of errors are recorded.
Change in Motor Inhibition after an exercise intervention | Change from baseline after 8 weeks
  Measured via cognitive tests on a computer screen using the ePrime software, which require participants to press a key on the keyboard every time a new image appears on the screen, except when a specific picture appears (specified in the instructions), in which case they must refrain from pressing the key. Reaction time (milliseconds) and number of errors are recorded.
Change in source memory after maximal exercise | Change from baseline after a single bout of maximal exercise (CPET)
  Measured via cognitive tests on a computer screen using the ePrime software, which require participants to recall specific details from an image shown previously. Reaction time (milliseconds) and number of errors are recorded.
Change in source memory after an exercise intervention | Change from baseline after 8 weeks
  Measured via cognitive tests on a computer screen using the ePrime software, which require participants to recall specific details from an image shown previously. Reaction time (milliseconds) and number of errors are recorded.
Changes in blood flow in the prefrontal cortex after maximal exercise | Change from baseline after a single bout of maximal exercise (CPET)
  Changes in saturation of oxy- and de-oxygenated blood in the prefrontal cortex of the brain as measured by near infrared spectroscopy (fNIRS). These two signals are then combined into one measure by using the correlation-based signal improvement (CBSI) procedure.
Changes in blood flow in the prefrontal cortex after an exercise intervention | Change from baseline after 8 weeks
  Changes in saturation of oxy- and de-oxygenated blood in the prefrontal cortex of the brain as measured by near infrared spectroscopy (fNIRS). These two signals are then combined into one measure by using the correlation-based signal improvement (CBSI) procedure.
Cognitive failures | Change from baseline after 8 weeks
  Measures via cognitive failures questionnaire. The questionnaire gives a score from 0-100, where a high number shows poor cognitive function.
Gum inflammation (oral health) | Baseline
  visual assessment of inflammation of the gum edge and measurement of the depth of the gum pocket (mm) following gentle probing with a calibrated blunt probe
Change in levels of Occupational Stress | Change from baseline after 8 weeks
  measured via Operational Police Stress Questionnaire (PSQ-Op),participants score 20 questions on a scale of 1-7, where 1 is no stress t alland 7 is very high stress.
Change in levels of Trauma | Change from baseline after 8 weeks
  measured via Impact of Events Scale (IES-R) questionnaires. Scores range from 0 - 88, where 0 is no trauma and 88 is severe trauma. A score of 24 or more signifies that PTSD is a clinical concern. 33 and above represents the best cutoff for a probable diagnosis of PTSD.
Change in Lifestyle - Physical activity levels | Change from baseline after 8 weeks
  Levels of physical activity measured via accelerometers and heart rate monitors using actigraphy, processed through the Actilife software. The software uses the two wearable devices to calculate proportions of the day spent in sedentary, light, moderate and vigorous activity. These measures are combined to show percentage of the day spent in each activity level.
Changes in Quality of Sleep (objective) | Change from baseline after 8 weeks
  Measured via accelerometers and heart rate monitors through Actilife software, which combined the heart rate and movement data from the wearable devices, providing a Sleep Efficiency score, reported as a percentage. A high percentage denotes good quality of sleep.
Changes in Quality of Sleep (subjective) | Change from baseline after 8 weeks
  Measured via and Pittsburg Sleep Quality Index (PSQI). The scale includes 7 items, each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Changes in Systemic inflammation | Change from baseline after 8 weeks
  hsCRP via Eurolyser
Changes in Risk of type II diabetes | Change from baseline after 8 weeks
  HBa1c via Eurolyser
Nutrition | Change from baseline after 8 weeks
  Eating habits assessed vi a Food Frequency Questionnaire, administered via an interview

CONTACTS AND LOCATIONS:
Locations (1):
- The ISEH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be anonymised and will be reported as group mean data